CLINICAL TRIAL: NCT02806921
Title: Protease and Cytokine Composition in Post Lens Tear Reservoir of Scleral Lenses for Keratoconic Eyes
Brief Title: Changes in the Tear Film With Scleral Contact Lens Wear for Keratoconic Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Principal Investigator, Luigina Sorbara, Associate Professor, University of Waterloo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 14620
Record Dates: First submitted 2016-06-16; First posted 2016-06-21 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Keratoconus
Keywords: Scleral Contact Lens; Tear Proteases; Tear Cytokines
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZenLens with Low limbal clearance (Active Comparator): Scleral contact lens designed to provide approximately 25 microns of limbal clearance.
  Interventions: Device: ZenLens
- ZenLens with High limbal clearance (Active Comparator): Scleral contact lens designed to provide approximately 80 microns of limbal clearance.
  Interventions: Device: ZenLens

INTERVENTIONS:
Device: ZenLens — The ZenLens™ semi-scleral lenses are manufactured by Alden Optic Laboratories Inc., Lancaster, NY. They will be made in Boston XO material.

SUMMARY:
The purpose of this study is to investigate changes in the level of inflammatory mediators in the tear film of scleral contact lens wearers in a keratoconic population.

DETAILED DESCRIPTION:
Scleral contact lenses are rigid gas permeable lenses designed to rest on the sclera while vaulting over the cornea with a fluid reservoir. The use of scleral contact lenses has become the current standard of practice as a nonsurgical management of corneal ectasia and ocular surface diseases. Cases have been recently presented of scleral lens wearers exhibiting adverse corneal findings and conjunctival injection from lens wear. These findings are likely associated with the mechanical and hypoxic effects due to poor fitting characteristics at the limbal area. Tear film analysis detecting changes in the levels of proteinases and cytokines have helped researchers gain a better understanding of the pathophysiology of complications in soft contact lenses wearers, dry eye, and keratoconus. Ultimately, this study will provide insights in relating scleral lens fitting characteristics and corneal and limbal physiological responses.

ELIGIBILITY:
Inclusion Criteria:

* Had been diagnosed with keratoconus in at least one eye.
* Is at least 18 years of age and has full legal capacity to volunteer.
* Has read and understood the information consent letter.
* Is willing and able to follow instructions and maintain the appointment schedule.

Exclusion Criteria:

* Is using any topical medications that will affect ocular health.
* Has any ocular pathology or severe insufficiency of lacrimal secretion (severe dry eyes) that would affect the wearing of contact lenses.
* Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye.
* Has any clinically significant lid or conjunctival abnormalities and active neovascularization.
* Is aphakic.
* Has undergone any corneal surgery.
* Is participating in any other type of eye related clinical or research study.
* Has any known allergies or sensitivity to the diagnostic pharmaceuticals or products, such as fluorescein, used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Tear Protein | 2 weeks of lens wear with daily schedule of 6-8 hours.
  To measure the level proteases and cytokines in each of the samples using Meso Scale Discovery system (MSD-ECL).

SECONDARY OUTCOMES:
Comfort | 2 weeks of lens wear with daily schedule of 6-8 hours.
  Participants will be asked to rate their ocular comfort, dryness, burning and vision with the contact lenses.
Bulbar and limbal hyperemia | 2 weeks of lens wear with daily schedule of 6-8 hours.
  The eyes of the participants will be imaged using the Keratograph® 5.
Corneal thickness | 2 weeks of lens wear with daily schedule of 6-8 hours.
  Their corneal thickness will be measured with the Visante OCT.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Informed Consent Form (2016-06-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT02806921/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-02-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT02806921/Prot_SAP_001.pdf